CLINICAL TRIAL: NCT02571192
Title: A Phase 1, Open-label Study to Investigate the Absorption, Distribution, Metabolism, and Excretion of [14C]-SHP626 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study to Investigate How the Study Drug SHP626 is Eliminated From the Body After One Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHP626-102
Record Dates: First submitted 2015-09-30; First posted 2015-10-08 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: ADME
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — volixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Drug (Experimental): single oral dose radiolabelled 50mg of SHP626
  Interventions: Drug: SHP626; Radiation: 5.95 μCi RAD

INTERVENTIONS:
Drug: SHP626 — single oral dose 50mg SHP626 with approximately 5.95 μCi RAD
Radiation: 5.95 μCi RAD

SUMMARY:
The purpose of this study is to determine how SHP626 is absorbed and excreted from the body in healthy males.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years, inclusive, at the time of consent.
2. Must be considered healthy. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, thyroid panel (includes T3, T4 and TSH at Screening only), blood chemistry, coagulation and urinalysis
3. Must have a body mass index between 18.0-30.0kg/m² inclusive with a body weight >50 kg (110 lbs).
4. Ability to swallow all investigational product.
5. A minimum of 1 bowel movement per day.

Exclusion Criteria:

1. History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gallbladder removal, gastric bypass surgery, ileal resection, any small intestinal resection,or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
2. Current or relevant history of physical or psychiatric illness.
3. Known or suspected intolerance or hypersensitivity to the investigational product, or closely-related compounds, or any of the stated ingredients.
4. Significant illness, as judged by the investigator, within 2 weeks of the dose of investigational product.
5. Known history of alcohol or other substance abuse within the last year.
6. Donation of blood or blood products (eg, plasma or platelets) within 60 days prior to the dose of investigational product.
7. Within 30 days prior to the dose of investigational product:

   * Have used an investigational product (if elimination half-life is <6 days, otherwise 5 half-lives).
   * Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.
   * Have had any substantial changes in eating habits, as assessed by the investigator.
8. Confirmed systolic blood pressure >139mmHg or <89mmHg, and diastolic blood pressure >89mmHg or <49mmHg.
9. Twelve-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450msec, the ECG should be repeated 2 more times and the average of the 3 QTc values should be used to determine the subject's eligibility.
10. A positive screen for drugs of abuse at Screening or a positive screen for alcohol or drugs of abuse at Check-in (Day -1).
11. Male subjects who consume more than 21 units of alcohol per week or 3 units of alcohol per day.
12. A positive human immunodeficiency virus antibody screen, hepatitis B surface antigen, or hepatitis C virus antibody screen.
13. Use of tobacco in any form
14. Routine consumption of more than 2 units of caffeine per day
15. Current use of any medication including over-the-counter, herbal, or homeopathic preparations
16. An inability to follow a standardized diet and meal schedule or inability to fast
17. Have participated in a [14C]-study within the last 6 months prior to the dose of investigational product.
18. Exposure to clinically significant radiation within 12 months prior to the dose of investigational product

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10-01; Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters will be determined from the plasma and blood concentration time data of total radioactivity and from the plasma concentration-time data for SHP626 by non-compartmental analysis. | Day 1 to day 10
Total radioactivity (RAD) in whole blood and plasma | Day 1 to day 10
To determine the total RAD in urine and feces. | Day 1 to day 10
Maximum plasma concentration (Cmax) of 50mg [14C]-SHP626 and RAD occurring at time of maximum observed concentration (tmax) | Day 1 to day 10
Area under the plasma concentration curve (AUC0-t) of 50mg [14C]-SHP626 and RAD from the time of dosing to the last measurable concentration | Day 1 to Day 10
Area under the plasma concentration curve (AUC0-∞ ) of 50mg [14C]-SHP626 and RAD extrapolated to infinity, calculated using the observed value of the last non-zero plasma concentration | Day 1 to Day 10
First order rate constant associated with the terminal portion of the plasma curve terminal half-life (t½) for 50mg [14C]-SHP626 and RAD | Day 1 to Day 10
Total body clearance (CL/F ) of 50mg [14C]-SHP626 and RAD for extravascular administration divided by the fraction of dose absorbed | Day 1-10
Volume of distribution (Vz/F ) of 50mg [14C]-SHP626 and RAD associated with the terminal slope following extra-vascular administration divided by the fraction of dose absorbed | Day 1-10
Cumulative amount (Aef )of RAD recovered in stool over the dosing interval | Day 1-10
Excreted Percent of RAD recovered in stool over the dosing interval | Day 1-10
Cumulative amount (Aeu ) of RAD recovered in urine over the dosing interval | Day 1-10
Excreted Percent of RAD recovered in urine over the dosing interval | Day 1-10
Renal Clearance (CLR ) of 50mg [14C]-SHP626 | Day 1 -10

SECONDARY OUTCOMES:
Characterize and identify metabolites of [14C]-SHP626 in plasma by accelerator mass spectrometry for radioactivity quantification | Day 1 to day 10
  Metabolites in the excreta and/or plasma will then be structurally identified by a combination of techniques such as co-chromatography with authentic reference standards, high performance liquid chromatography-mass spectrometry, and other spectroscopic techniques if necessary
Characterize and identify metabolites of [14C]-SHP626 in urine by accelerator mass spectrometry for radioactivity quantification | Day 1 to day 10
  Metabolites in the excreta and/or plasma will then be structurally identified by a combination of techniques such as co-chromatography with authentic reference standards, high performance liquid chromatography-mass spectrometry, and other spectroscopic techniques if necessary
Characterize and identify metabolites of [14C]-SHP626 in feces by liquid scintillation counting | Day 1 to day 10
  Metabolites in the excreta and/or plasma will then be structurally identified by a combination of techniques such as co-chromatography with authentic reference standards, high performance liquid chromatography-mass spectrometry, and other spectroscopic techniques if necessary
Assess the safety and tolerability of [14C]-SHP626 by adverse events (AEs) defined as changes, including changes from baseline in physical examination findings | Screening to day 7
  AEs will be coded using the agreed upon version of MedDRA. The number of events, incidence, and percentage of TEAEs will be calculated overall, by system organ class and by preferred term. TEAEs will be further summarized by severity and relationship to investigational product. AEs related to investigational product, AEs leading to withdrawal, SAEs, and deaths will be similarly summarized/listed.
Changes from baseline in vital signs | Screening to day 7
Changes from baseline in ECGs | Screening to day 7
Changes from baseline in hematology | Screening to day 7
Changes from baseline in coagulation | Screening to day 7
Changes in baseline in urinalysis | Screening to day 7
Changes in baseline in chemistry | Screening to day 7

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, MD, Principal Investigator — Covance Clinical Pharmacology
Locations (1):
- Covance Madison Clinical Research Unit, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Siebers N, Palmer M, Silberg DG, Jennings L, Bliss C, Martin PT. Absorption, Distribution, Metabolism, and Excretion of [14C]-Volixibat in Healthy Men: Phase 1 Open-Label Study. Eur J Drug Metab Pharmacokinet. 2018 Feb;43(1):91-101. doi: 10.1007/s13318-017-0429-7. PMID 28702877